CLINICAL TRIAL: NCT02443727
Title: The Role of Oxytocin in the Perception of Infant Faces
Brief Title: The Role of Oxytocin in the Perception of Faces
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Rodrigo Cardenas (Other)
Collaborators: U.S. National Science Foundation (U.S. Federal Agency)
Responsible Party: Sponsor-Investigator, Rodrigo Cardenas, Lecturer, Penn State University
Organization: Penn State University (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: STUDY00001225
Record Dates: First submitted 2015-05-05; First posted 2015-05-14 (Estimated); Last update posted 2023-04-25 (Actual); Status verified 2023-04

CONDITIONS: Healthy
MeSH Terms: interventions — Oxytocin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Intranasal oxytocin group (Experimental): Participants will self-administer a single dose of 24 IU oxytocin (Syntocinon, Novartis; three puffs per nostril, each with 4 IU oxytocin, 6 puffs total).
  Interventions: Drug: Syntocinon (synthetic oxytocin)
- Placebo group (Placebo Comparator): The placebo is identical to the oxytocin formulation with the exception of the active compound.
  Participants will self-administer three puffs per nostril of placebo (6 puffs total).
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Syntocinon (synthetic oxytocin) — Dosage and details described in arm.
  Other Names: OT
  Arms: Intranasal oxytocin group
Other: Placebo — Dosage and details described in arm.
  Arms: Placebo group

SUMMARY:
The main objective of this project is to study whether intranasal oxytocin (OT) affects how young adults perceive and attend to infant and adult faces. Based on existing research the investigators predict that oxytocin will facilitate the allocation of attentional resources on infant faces (compared to adult faces). The investigators also predict that oxytocin will enhance the activity of reward neural-networks associated with the perception of infant faces. The behavioral effects of OT (visual attention and face recognition) will be measured with eye-tracking while participants look at photographs of adult and infant faces. Neurological effects (the activity of emotion and reward networks) will be measured with functional Magnetic Resonance Imaging (fMRI) while participants look at infant faces on a computer screen.

ELIGIBILITY:
Inclusion Criteria:

* Healthy Volunteers
* Norma or corrected to norma vision
* Participants are non parents
* Able to provide written informed consent and to comply with all study procedures

Exclusion Criteria:

* Dementia or severe cognitive disorders
* Endocrine disease or malignancy
* Nasal obstruction or upper-respiratory tract infection
* Current or previous psychiatric disorder
* Current or previous use of psychoactive drugs
* Alcoholism or substance abuse
* History of seizures
* Neurological Disorder
* Previous head trauma
* Hypertension
* Cardiovascular Disease
* Claustrophobia
* ferrous metal in any part of the body

Ages: 18 Years to 25 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 71 (Actual)
Dates: Start 2015-04 (Actual); Primary Completion 2015-12 (Actual); Study Completion 2016-09 (Actual)

PRIMARY OUTCOMES:
Functional Magnetic Resonance Imaging (fMRI) Data | 45 minutes after OT manipulation
  The effect of OT will be assessed by determining changes in brain activation between treatment and placebo groups.
Eye movements data | 45 minutes after OT manipulation
  The effect of OT will be assessed by determining changes in eye movements between treatment and placebo groups.

SECONDARY OUTCOMES:
Implicit Attitudes toward infants | 45 minutes after OT manipulation
  Implicit attitudes toward infants as measured by the Implicit Association Test
Theory of mind | 45 minutes after OT manipulation
  Theory of mind as measured by the Reading the mind in the eyes test

CONTACTS AND LOCATIONS:
Overall Officials: Rodrigo A Cardenas, PhD, Principal Investigator — Penn State University